CLINICAL TRIAL: NCT06874608
Title: Evaluation of the Efficacy and Tolerability of an Exclusion Diet in Patients With Juvenile Idiopathic Arthritis: Interventional, Exploratory Single-center, Randomized, Controlled, Open-label, add-on Study
Brief Title: Evaluation of the Efficacy and Tolerability of an Exclusion Diet in Patients With Juvenile Idiopathic Arthritis
Acronym: JIA-ED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Paolo Lionetti, Principal Investigator, Meyer Children's Hospital IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: JIA-ED
Record Dates: First submitted 2025-02-25; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Juvenile Idiopathic Arthritis (JIA)
Keywords: JIA; CDED; Dietary therapy
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Dietary Fiber; Lactose; Diet, Gluten-Free

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): In this arm patients of newly diagnosis, or who failed synthetic or biologic therapy will be treated with standard of care therapy and free diet
- Intervention arm (Experimental): In this arm patients of newly diagnosis, or who failed synthetic or biologic therapy will be treated with the Crohn Disease Exclusion Diet (CDED) plus partial enteral nutrition
  Interventions: Dietary Supplement: complete, polymeric formula, fiber, lactose and gluten free

INTERVENTIONS:
Dietary Supplement: complete, polymeric formula, fiber, lactose and gluten free — The dietary intervention attempts to induce remission in the first 4-week treatment without any change in the pharmaceutical therapy. In case of worsening or not reaching the outcomes, the patient will be defined as a failure and start rescue therapy with the standard of care.
  Arms: Intervention arm

SUMMARY:
The JIA-ED study is a pilot project. Based on experience in another inflammatory disease, a 4-week period was extrapolated as sufficient to assess the effectiveness of the experimental intervention. This observation is supported by literature data showing that, halfway through phase I of the CDED (Crohn Diseasse Exclusion Diet), it is already possible to identify a subset of patients with Crohn's disease who are responsive to the dietary treatment and who also have a higher likelihood of achieving clinical remission by the end of the first phase of the diet itself.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of juvenile idiopathic arthritis (JIA) in the forms of enthesitis-related arthritis and oligoarticular forms according to the ILAR 2001 criteria (https://medicalcriteria.com/web/reujia/);
* Age between 6 and 18 years (not yet 18);
* Active disease of mild to moderate severity, assessed through the Juvenile - Arthritis Disease Activity Score (JADAS10) tool (Trincianti C. et al., American College Rheumatology, 2021);
* For study groups 2 and 3: failure of ongoing pharmacological therapy at the time of screening, defined as a failure to achieve at least a 20% reduction in JADAS10 values after 3 months of initiating DMARD therapy or biologic medication, or if the disease is inactive on such therapy, a 20% increase in those values;
* Signed informed consent.

Exclusion Criteria:

* Patients requiring systemic immunosuppressive therapy for active uveitis;
* Patients undergoing therapy with systemic corticosteroids (defined as prednisone equivalent >0.5 mg/kg for >7 days) or intra-articular corticosteroids in the 3 months prior to enrollment;
* Patients with fecal calprotectin values > 250 mcg/g at the time of screening;
* Use of antibiotics in the month prior to enrollment.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Number of patients showing 20% improvement in juvenile arthritic disease activity score (JADAS) | Baseline, 4 weeks, 8 weeks post-enrollment

SECONDARY OUTCOMES:
Number of patients showing a high score on the Modulence Adherence Rating Scale (MARS) | Week 4, week 8, week 16, week 26 post-enrollment
Number of patients showing reduction of Reactive C Protein (RCP) after exclusion diet | Baseline, 4 weeks, 8 weeks post-enrollment
Number of patients showing reduction of erythrocyte sedimentation rate (ESR) after exclusion diet | Baseline, 4 weeks, 8 weeks post-enrollment

OTHER OUTCOMES:
Percentage of patients with gut microbiota modifications | Baseline, week 4, week 8, week 16, week 26 post-enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Meyer IRCCS, Florence, Italy

IPD SHARING:
Plan to Share IPD: No